CLINICAL TRIAL: NCT03017144
Title: The Association Between Technical and Non-technical Skills in Real-life ALS Situations. Impact of Pit Crew Model on the Resuscitation Skills.
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T70/2012
Record Dates: First submitted 2016-10-17; First posted 2017-01-11 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Arrest
Keywords: non-technical skills (NTS); human factors; team work; Crew Resource Management / Crisis Resource Management (CRM); technical skills (TS); Cardiopulmonary resuscitation; Advanced cardiac life support; Pit Crew Model
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resuscitation team: Resuscitation pit crew model is educated to the resuscitation team.
  Interventions: Other: Pit crew model education

INTERVENTIONS:
Other: Pit crew model education — A pit crew model for resuscitation is educated to all resuscitation team members.

SUMMARY:
Cardiac arrest is handled by cardiopulmonary resuscitation which is a time critical emergency situation. The actions during resuscitation are lead by international guidelines. Traditionally, the main focus of the training has been on medical knowledge and technical skills (TS). Nowadays non-technical skills (NTS), such as communication, teamwork behaviour, and leadership, are considered at least equally important.

The aim of this study is to evaluate both TS and NTS of the resuscitation team during real-life resuscitation situations using a validated assessment tool. The association between TS and NTS will be analyzed. Findings from this study may help to recognize the possible weaknesses and issues which could be improved by training. Hypothesis is that that TS are probably in a high level, but some improvement points of NTS are ought to be known better. Investigators hypothesis that the good NTS performance in resuscitation is accompanied by good TS performance.

DETAILED DESCRIPTION:
Background

Cardiac arrest is a time-critical emergency situation, which is treated by cardiopulmonary resuscitation (CPR). The actions during resuscitation are lead by international guidelines (Nolan et al 2010). Because of the relatively rare nature of cardiac arrests in many wards and clinics, regular resuscitation training is necessary.

During cardiopulmonary resuscitation and other sudden medical crisis situations, in addition to medical knowledge and technical skills (TS), also non-technical skills (NTS) are needed (Castelao et al 2011, Fletcher et al 2002, Helmreich et al 1999, Gaba et al 1998). NTS are behavioural elements which are ought to improve team performance. The importance of NTS has been demonstrated only in a simulated settings, not in a real life.

Drawbacks in team organization and communication are frequent problems within advanced life support (ALS) events (Risaliti et al, Colquitt et al). As unclear team member roles can cause errors during ALS (Weng et al, Ornato et al) more emphasis should be placed on educating specific roles and responsibilities to resuscitation team members (Soar et al, Maney et al). Pit crew models for resuscitation, where all resuscitation team members have their pre-assigned positions and pre-arranged roles and tasks to perform ALS have been developed to respond these problems. (Gonzales et al, Pearson et al, Glendenning et al, Ong et al, Hopkins et al, Spitzer et al)

Objective, purpose, and hypothesis

The first part of this study (ID T70/2012) aims to evaluate the technical and especially non-technical skills of the resuscitation team during real-life resuscitation situations. Investigators hypothesis that good non-technical performance is related on good technical performance. Findings from this study may help to recognize the possible weaknesses and issues which could be improved by training. The hypothesis is that technical skills are probably on a high level, but some improvement points of non-technical skills are ought to be known better.

The second part of the study aims to evaluate the impact of a pit crew model on ALS skills. (ID: T70/2012)

Design and Methods

Turku University Central Hospital lies in a Southwestern part of Finland, and provides medical services for 865 000 inhabitants. The target group of this study is the resuscitation team of the adult ICU of Turku University Central Hospital. This team consists of an ICU doctor (most commonly an anaesthesiologist specialized for intensive care), two ICU nurses, and one medical technician. These people are treating approximately 90 cardiac arrests per year, but this group also gets other alarms (like shortness of breath, unconscious patients and other acute situations). This ICU resuscitation team takes care of all resuscitation calls in the newer part of the Turku University Hospital, when the older parts of the hospital are taken care either by a resuscitation team from pediatric ICU or by prehospital emergency medical service system.

The data from 20 video-recorded real-life resuscitation situations treated by resuscitation team in Turku University Hospital will be collected and the overall NTS and TS score will be measured using a validated assessment tool (Peltonen et al 2017). The association between the TS and NTS will be analyzed by statistical methods. In addition, after each recorded resuscitation situation, every member of the resuscitation team will be called by a phone. During the calls team members are asked to tell examples, what went well during the resuscitation, and what could have been done better. Based on these answers, inductive analysis will be made.

A pit crew model for resuscitation will be implemented in our organizations' resuscitation team responding cardiac arrest alarms. We will continue to video-recording after the intervention, and similarly, NTS and TS will be measured using the validated assessment tool (Peltonen et al 2017). In the second part of the study, we will compare the pre- and post-intervention ALS-performance in the videos.

Ethics

The study protocol was approved by the Ethics Committee of Turku University. All ALS-situations in Turku University newer hospital building area are considered eligible to the study regardless of the initial rhythm or presumed aetiology. Written information consent of patients is not needed, because the study is directed at resuscitation team performance, not the patients. The patients are not identified at any phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. a doctor, a nurse, a paramedic or a medical technician working on adult ICU resuscitation team
2. all the members of the ICU resuscitation team in the CPR-situation are volunteer to take part in the study

Exclusion Criteria:

1) if any member of the ICU resuscitation team in the CPR-situation refuse to be video recoded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target group of this study is the resuscitation team of the adult ICU of Turku University Central Hospital. This team consists of an ICU doctor (most commonly an anaesthesiologist specialized for intensive care), two ICU nurses and one medical technician.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
To measure the association of the NTS and TS on one-another using validated assessment tool. | one year

SECONDARY OUTCOMES:
To evaluate the association between NTS and TS subgategories. | one year

OTHER OUTCOMES:
To evaluate the impact of the pit crew model in the second part of the study. | two years
  The primary outcome will be the difference in TS and NTS total scores pre- and post intervention. Secondary outcome will be the diccerence in TS and NTS subcategories and hands-on-time.

CONTACTS AND LOCATIONS:
Overall Officials: Miretta Tommila, MD, Principal Investigator — Turku University Hospital; Sanna Salanterä, PhD, RN, Study Director — Vice Head of the Department of Nursing Science and Nurse Director at Turku University Hospital, Finland; Ville Peltonen, Lic.Med, Study Chair — Turku University Hospital; Laura-Maria Peltonen, M.Sc. RN, Study Chair — University of Turku, Finland, Nursing Science; Teemu Elomaa, Lic.Med, Study Chair — Turku University Hospital; Jaana Elomaa, RN, Study Chair — Turku University Hospital; Tomi Pappila, RN, Study Chair — Vakka-Suomi Hospital Tyks, Finland; Sanna Hoppu, MD, Study Chair — Tampere University Hospital, Finland; Eeva Hevonoja, RN, Study Chair — University of Turku, Finland; Saija Hurme, Study Chair — University of Turku, Finland; Katariina Perkonoja, Study Chair — University of Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Patients treated by cardiopulmonary resuscitation (CPR) in the videos can be recognized. Video material can not be shared due to patient privacy. Other data is possible to share.

REFERENCES:
- [Background] Nolan JP, Soar J, Zideman DA, Biarent D, Bossaert LL, Deakin C, Koster RW, Wyllie J, Bottiger B; ERC Guidelines Writing Group. European Resuscitation Council Guidelines for Resuscitation 2010 Section 1. Executive summary. Resuscitation. 2010 Oct;81(10):1219-76. doi: 10.1016/j.resuscitation.2010.08.021. No abstract available. PMID 20956052
- [Background] Fernandez Castelao E, Russo SG, Cremer S, Strack M, Kaminski L, Eich C, Timmermann A, Boos M. Positive impact of crisis resource management training on no-flow time and team member verbalisations during simulated cardiopulmonary resuscitation: a randomised controlled trial. Resuscitation. 2011 Oct;82(10):1338-43. doi: 10.1016/j.resuscitation.2011.05.009. Epub 2011 May 25. PMID 21664757
- [Background] Fletcher GC, McGeorge P, Flin RH, Glavin RJ, Maran NJ. The role of non-technical skills in anaesthesia: a review of current literature. Br J Anaesth. 2002 Mar;88(3):418-29. doi: 10.1093/bja/88.3.418. No abstract available. PMID 11990277
- [Background] Helmreich RL, Merritt AC, Wilhelm JA. The evolution of Crew Resource Management training in commercial aviation. Int J Aviat Psychol. 1999;9(1):19-32. doi: 10.1207/s15327108ijap0901_2. PMID 11541445
- [Background] Gaba DM, Howard SK, Flanagan B, Smith BE, Fish KJ, Botney R. Assessment of clinical performance during simulated crises using both technical and behavioral ratings. Anesthesiology. 1998 Jul;89(1):8-18. doi: 10.1097/00000542-199807000-00005. PMID 9667288
- [Derived] Peltonen V, Peltonen LM, Salantera S, Hoppu S, Elomaa J, Pappila T, Hevonoja E, Hurme S, Perkonoja K, Elomaa T, Tommila M. An observational study of technical and non-technical skills in advanced life support in the clinical setting. Resuscitation. 2020 Aug;153:162-168. doi: 10.1016/j.resuscitation.2020.06.010. Epub 2020 Jun 16. PMID 32561474